CLINICAL TRIAL: NCT03384277
Title: A Prospective, Randomized, Multicenter Clinical Trial of Acquired Haemophilia A With Steroid Combined With Cyclophosphamide Versus Steroid Combined With Rituximab
Brief Title: Trial of Acquired Haemophilia With Steroid Combined With Cyclophosphamide Versus Steroid Combined With Rituximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Tianjin First Central Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2017006
Record Dates: First submitted 2017-11-28; First posted 2017-12-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2023-06

CONDITIONS: Acquired Hemophilia A
Keywords: Acquired hemophilia A; Cyclophosphamide; Rituximab; Steroid
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Steroids; Adrenal Cortex Hormones; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid+Rituximab (Experimental): Methylprednisolone 0.8 mg/kg/day (or equivalent corticosteroid doses) for 3 weeks（then tapering gradually, 8 weeks in total）+Rituximab 375mg/m2 for one dose.
  Interventions: Drug: Steroid; Drug: Rituximab
- Steroid +Cyclophosphamide (Active Comparator): Methylprednisolone 0.8 mg/kg/day (or equivalent corticosteroid doses) for 3 weeks （ then tapering gradually, 8 weeks in total）+ Cyclophosphamide 2 mg/kg/day until inhibitor negative (no longer than five weeks)
  Interventions: Drug: Steroid; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Steroid — Methylprednisolone 0.8 mg/kg/day (or equivalent corticosteroid doses) for 3 weeks（then tapering gradually, 8 weeks in total）
  Other Names: Corticosteroid
Drug: Rituximab — 375mg/m2 for one dose
  Arms: Steroid+Rituximab
Drug: Cyclophosphamide — cyclophosphamide 2 mg/kg/day until inhibitor negative (no longer than five weeks)
  Arms: Steroid +Cyclophosphamide

SUMMARY:
Purpose:

To evaluate the efficacy when administering steroid combined with single dose rituximab to eliminate the antibody in acquired hemophilia A patients compared to treatment using steroid with cyclophosphamide.

The study will test the hypothesis that steroid combined with small dose rituximab is as effective as steroid combined with cyclophosphamide for FVIII inhibitor eradication in Chinese patients with acquired hemophilia A.

Study design Allocation: Randomized Intervention Model: Parallel Assignment Masking: None (Open Label) Primary Purpose: Treatment

DETAILED DESCRIPTION:
This is a prospective randomized multi-center controlled pilot trial comparing the regimen of steroid with rituximab and steroid with cyclophosphamide to eradicate anti-factor VIII antibodies in Chinese patients with acquired hemophilia A.

Patients will be randomized to two regimens: methylprednisolone 0.8mg/kg/day (or equivalent corticosteroid doses) for 3 weeks (then tapering gradually,8 weeks in total) with rituximab (375mg/m2 for one dose) or methylprednisolone 0.8mg/kg/day (or equivalent corticosteroid doses) for 3 weeks (then tapering gradually,8 weeks in total) with cyclophosphamide 2mg/kg/day until inhibitor negative(no longer than five weeks).

Patients will be randomized to the treatment cohorts according to the biostatistical methods.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Men or women
* Women post-menopausal or with ongoing contraception
* Diagnosis of acquired hemophilia A
* Patient must be insured
* Patient has provided written informed consent prior to enrollment
* Patient compliant

Exclusion Criteria:

* Congenital hemophilia
* Ongoing treatment with prednisone > 20mg/d （or equivalent corticosteroid doses） more than 1 month
* Ongoing treatment with prednisone >0.7mg/kg（or equivalent corticosteroid doses） more than 10 days
* Pregnant and breastfeeding women
* Allergy to steroid
* Immunosuppressive agents treatment within 30 days
* Serum transaminase and bilirubin greater than 1.5 times the upper limit of normal value
* Hepatitis B surface antigen or hepatitis C antibody or HIV antibody (I + II) or syphilis antibody positive
* Patients with diabetes, hypertension, glaucoma, peptic ulcer, herpes zoster, pulmonary infection and so on, who should not be treated with glucocorticoids
* Patients with poor compliance
* Those who can not take contraceptive measures during the test period
* Patient who is considered by the investigator not suitable for clinical study
* Thrombocytopenia
* Leucocytopenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Proportion of inhibitor eradication and time to attain first remission | During 18 months
  The proportion of patients achieving complete remission (CR) defined as titer FVIII inhibitor lower than 0.6 Bethesda unit, factor VIII level> 50% and no bleeding events without bypass treatments for 24 hours and the time to attain first remission will be evaluated.

SECONDARY OUTCOMES:
Relapse rate and time to relapse | During 18 month
  The proportion of patients who relapse and the time to relapse of each regimen will be measured.

OTHER OUTCOMES:
Infection of two regimens | During 18 months
  The safety outcomes will be the occurrence of infection related to immunosuppressive treatment adverse events.
Hemocytopenia of two regimens | During 18 month
  The safety outcomes will be the occurrence of Hemocytopenia related to immunosuppressive treatment adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Blood disease hospital, Chinese academy of medical sciences
Locations (1):
- Ethics Committee of Blood disease hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome will be made available
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available within 6 month of study completion
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requests will be required to sign a Data Access Agreement
URL: http://www.medresman.org

REFERENCES:
- [Background] Collins P, Baudo F, Huth-Kuhne A, Ingerslev J, Kessler CM, Castellano ME, Shima M, St-Louis J, Levesque H. Consensus recommendations for the diagnosis and treatment of acquired hemophilia A. BMC Res Notes. 2010 Jun 7;3:161. doi: 10.1186/1756-0500-3-161. PMID 20529258
- [Background] Collins PW, Hirsch S, Baglin TP, Dolan G, Hanley J, Makris M, Keeling DM, Liesner R, Brown SA, Hay CR; UK Haemophilia Centre Doctors' Organisation. Acquired hemophilia A in the United Kingdom: a 2-year national surveillance study by the United Kingdom Haemophilia Centre Doctors' Organisation. Blood. 2007 Mar 1;109(5):1870-7. doi: 10.1182/blood-2006-06-029850. Epub 2006 Oct 17. PMID 17047148
- [Background] Lottenberg R, Kentro TB, Kitchens CS. Acquired hemophilia. A natural history study of 16 patients with factor VIII inhibitors receiving little or no therapy. Arch Intern Med. 1987 Jun;147(6):1077-81. doi: 10.1001/archinte.147.6.1077. PMID 3109341
- [Background] Collins P, Baudo F, Knoebl P, Levesque H, Nemes L, Pellegrini F, Marco P, Tengborn L, Huth-Kuhne A; EACH2 registry collaborators. Immunosuppression for acquired hemophilia A: results from the European Acquired Haemophilia Registry (EACH2). Blood. 2012 Jul 5;120(1):47-55. doi: 10.1182/blood-2012-02-409185. Epub 2012 Apr 18. PMID 22517903
- [Background] Stasi R, Brunetti M, Stipa E, Amadori S. Selective B-cell depletion with rituximab for the treatment of patients with acquired hemophilia. Blood. 2004 Jun 15;103(12):4424-8. doi: 10.1182/blood-2003-11-4075. Epub 2004 Mar 2. PMID 14996701
- [Derived] Wang P, Zhou R, Xue F, Zhou H, Bai J, Wang X, Ma Y, Song Z, Chen Y, Liu X, Fu R, Sun T, Ju M, Dai X, Dong H, Yang R, Liu W, Zhang L. Single-dose rituximab plus glucocorticoid versus cyclophosphamide plus glucocorticoid in patients with newly diagnosed acquired hemophilia A: A multicenter, open-label, randomized noninferiority trial. Am J Hematol. 2024 Jan;99(1):28-37. doi: 10.1002/ajh.27128. Epub 2023 Oct 18. PMID 37851608